CLINICAL TRIAL: NCT05829278
Title: Efficacy and Central Mechanism of Acupuncture for Treating Chronic Subjective Tinnitus Assessed by fNIRS: Study Protocol for a Randomized Controlled Pilot Trial
Brief Title: Efficacy and Central Mechanism of Acupuncture for Treating Chronic Subjective Tinnitus Assessed by fNIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Hantong Hu, Principal Investigator, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YLKY-2021-01-01
Record Dates: First submitted 2023-04-11; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Tinnitus
Keywords: acupuncture; moxibustion; tinnitus; randomized controlled trial
MeSH Terms: conditions — Tinnitus | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Subjects in the acupuncture group will undergo acupuncture treatment, which is administered 3 times a week for 4 weeks.
  Interventions: Procedure: Acupuncture
- Waiting list group (No Intervention): No intervention will be provided for the waiting list group and the subjects in this group will be followed during the 4-week observation period.

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture will be performed at acupoints including TE17 (Yifeng), SI19 (Tinggong), GB2 (Tinghui), TE5 (Waiguan), TE3 (Zhongzhu), ST36(Zusanli ), KI3 (Taixi), and etc.
  Arms: Acupuncture group

SUMMARY:
This randomized controlled pilot trial aims to explore the Efficacy and central mechanism of acupuncture for treating chronic subjective tinnitus using functional near-infrared spectroscopy (fNIRS).

DETAILED DESCRIPTION:
A total of 60 tinnitus patients were randomly assigned to either an acupuncture group or a waiting list group in a 1:1 ratio. Subjects in the acupuncture group will undergo 4-week acupuncture treatment, while subjects in the waiting list group will receive no treatment during the 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral tinnitus that meets the diagnostic criteria for chronic subjective tinnitus.
2. Male and female, Aged between 18 and 60 years.
3. Participants can cooperate with experimental procedures and sign written inform consent.
4. Not participating in other clinical trials concurrently.

Exclusion Criteria:

1. Participants with objective tinnitus
2. Participants have nervous system diseases or neuropsychiatric diseases that can significantly affect brain blood oxygen metabolism assessed by resting-state functional connectivity.
3. Participants with severe cardiovascular and cerebrovascular diseases, malignant liver and kidney diseases, and other serious diseases.
4. Participants have any contraindications for acupuncture (such as a bleeding tendency)
5. Pregnant or lactating women.
6. Participants have received tinnitus treatment with drugs or other therapies in the last four weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in resting-state functional connectivity (RSFC) | at baseline (pre-treatment), at 4 weeks after intervention, at 3-month follow-up
  RSFC will be measured by functional near-infrared spectroscopy (fNIRS).
Change in hemoglobin signals | at baseline (pre-treatment), at 4 weeks after intervention, at 3-month follow-up
  Hemoglobin signals will be measured by functional near-infrared spectroscopy (fNIRS).

SECONDARY OUTCOMES:
Change in Tinnitus Handicap Inventory score | at baseline (pre-treatment), at 4 weeks after intervention, at 3-month follow-up
  Tinnitus Handicap Inventory contains 25 items, each valued at 0-4 points. A larger score indicates a more severe degree of tinnitus.
Change in average pure-tone threshold | at baseline (pre-treatment), at 4 weeks after intervention, at 3-month follow-up
  Average pure-tone threshold will be assessed by pure-tone audiometry.
Change in Hamilton Anxiety Scale score | at baseline (pre-treatment), at 4 weeks after intervention, at 3-month follow-up
  Hamilton Anxiety Scale is a reliable indicator of the severity of anxiety symptoms. The Hamilton Anxiety Scale consists of 14 items, each rated on a 5-point scale from 0 to 4. A larger score indicates a more severe degree of anxiety.
Change in tinnitus loudness | at baseline (pre-treatment), at 4 weeks after intervention, at 3-month follow-up
  Tinnitus loudness will be measure by using an 11-point numerical rating scale, with 0 indicating no tinnitus and 10 indicating maximum intolerable tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: Hantong Hu, M.D., Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuzucu I, Karaca O. Acupuncture Treatment in Patients with Chronic Subjective Tinnitus: A Prospective, Randomized Study. Med Acupunct. 2020 Feb 1;32(1):24-28. doi: 10.1089/acu.2019.1367. Epub 2020 Feb 3. PMID 32104524
- [Derived] Hu H, Lin X, Fang L, Li Y, Gao H. Evaluating the Efficacy and Underlying Mechanisms of Acupuncture for Chronic Subjective Tinnitus Using Functional Near-Infrared Spectroscopy: Study Protocol for a Randomized Controlled Trial. J Pain Res. 2023 Oct 4;16:3367-3378. doi: 10.2147/JPR.S433048. eCollection 2023. PMID 37814607